CLINICAL TRIAL: NCT01338480
Title: Improving Informed Consent Process for Trauma Patients in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Ko Lin, Attending Physician, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUH-IRB-980361
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Trauma; Surgery
Keywords: trauma; surgery; informed consent
MeSH Terms: conditions — Wounds and Injuries | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- video (Experimental): Participants in the intervention group watched an educational video illustrating informed consent information
  Interventions: Other: video
- control (No Intervention): Participants in the control group read an informed consent document.

INTERVENTIONS:
Other: video — The videos will be developed and contain information on the procedure, risks, benefits, and alternatives of the surgery. The knowledge measure instrument will also be developed.
  Arms: video

SUMMARY:
This study is planning to develop the audiovisual videos and determine whether educational videos are superior to routine discussion for informing trauma patients in emergency department (ED) about risks, benefits, and alternatives to receiving surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* scheduled to receive the surgery

Exclusion Criteria:

* clinically unstable
* refuse to participate
* unable to understand the consent process for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2009-11-09 (Actual); Primary Completion 2014-10-22 (Actual); Study Completion 2014-10-22 (Actual)

PRIMARY OUTCOMES:
knowledge score | immediately after the intervention
  The primary outcome, patient understanding of the procedure, risks, benefits, and alternatives, will be determined by quantitative scores on the written examination

SECONDARY OUTCOMES:
satisfaction | immediately after the intervention
  Secondary outcomes include patient satisfaction with the informed consent process, determined by a five-point ordinal satisfaction scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Ko Lin, M.D., Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan, Taiwan

REFERENCES:
- [Derived] Lin YK, Chen CW, Lee WC, Cheng YC, Lin TY, Lin CJ, Shi L, Tien YC, Kuo LC. Educational video-assisted versus conventional informed consent for trauma-related debridement surgery: a parallel group randomized controlled trial. BMC Med Ethics. 2018 Mar 9;19(1):23. doi: 10.1186/s12910-018-0264-7. PMID 29523129
- [Derived] Lin YK, Chen CW, Lee WC, Lin TY, Kuo LC, Lin CJ, Shi L, Tien YC, Cheng YC. Development and pilot testing of an informed consent video for patients with limb trauma prior to debridement surgery using a modified Delphi technique. BMC Med Ethics. 2017 Nov 29;18(1):67. doi: 10.1186/s12910-017-0228-3. PMID 29187226